CLINICAL TRIAL: NCT03872362
Title: Radiomics and Clinical Variables Can Differentiate Malignant Nodules and Detect Invasive Adenocarcinoma in Pulmonary Nodules: a Multi-center Study
Brief Title: Radiomics Multifactorial Biomarker for Pulmonary Nodules
Acronym: RMBPN
Status: Completed | Type: Observational
Sponsor: Maastricht University (Other)
Collaborators: Affiliated Zhongshan Hospital of Dalian University (Other); The Second Affiliated Hospital of Dalian Medical University (Other); The Fifth Hospital of Dalian (Unknown)
Responsible Party: Sponsor
Other Study IDs: UM2019DLABGY1
Record Dates: First submitted 2019-03-11; First posted 2019-03-13 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-01

CONDITIONS: Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Lung Diseases; Neoplasms; Pathology
Keywords: Lung cancer; CT; Frozen sections; Radiomics; Lung adenocarcinoma
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Lung Diseases; Neoplasms; Adenocarcinoma of Lung | interventions — Radiomics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Training dataset: No interventions
  Interventions: Diagnostic Test: radiomics
- External validation1: No interventions
  Interventions: Diagnostic Test: radiomics
- External validation2: No interventions
  Interventions: Diagnostic Test: radiomics

INTERVENTIONS:
Diagnostic Test: radiomics — The high-throughput extraction of large amounts of quantitative image features from medical images

SUMMARY:
The investigators aim to investigate the utility of radiomics to differentiate malignant nodules from benign nodules and invasive adenocarcinoma from non-invasive adenocarcinoma.

DETAILED DESCRIPTION:
With the development of computed tomography (CT) equipment and the increasing use of lung cancer screening programs with low-dose CT, a growing number of early-stage lung cancers were detected so that a large number of patients have undergone surgery.

Although a number of radiological studies have been used morphological signs so-called semantic features to make a differential diagnosis, it is still hard to apply by clinician because pulmonary nodules especially ground-glass nodules and small size nodules have atypical radiology signs and have strong subjectivity from different observers. Recently, CT-based radiomics, extracting the quantitative high-throughput features from medical images and facilitating clinical decision-making system, showed a good performance to predict diagnosis and prognosis of diverse cancer.

Therefore, the proposed project aims to develop and validate radiomics models based on CT images to identify malignant nodules and then to discriminate the different types of lung adenocarcinoma in patients with pulmonary nodules.

ELIGIBILITY:
Inclusion Criteria:

* intraoperative frozen section diagnosis and final pathology diagnosis are available
* preoperative standard non-enhanced CT is available
* Pathologically confirmed

Exclusion Criteria:

* with a previous history of radiation therapy, chemotherapy or biopsy
* the time interval between the CT examination and surgery was more than two weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pulmonary nodules in the collaborating institutes.
Sampling Method: Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2018-07-11 (Actual); Primary Completion 2019-01-11 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Malignant nodules classifier | 30 days
  Model based on Radiomic that can differentiate malignant nodules from benign nodules.
Invasive adenocarcinoma classifier | 30 days
  Model based on Radiomic that can differentiate invasive adenocarcinoma from non-invasive adenocarcinoma.

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Zhongshan Hospital of Dalian University, Dalian, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wu G, Woodruff HC, Shen J, Refaee T, Sanduleanu S, Ibrahim A, Leijenaar RTH, Wang R, Xiong J, Bian J, Wu J, Lambin P. Diagnosis of Invasive Lung Adenocarcinoma Based on Chest CT Radiomic Features of Part-Solid Pulmonary Nodules: A Multicenter Study. Radiology. 2020 Nov;297(2):451-458. doi: 10.1148/radiol.2020192431. Epub 2020 Aug 25. PMID 32840472